CLINICAL TRIAL: NCT06955689
Title: Effectiveness of the Localized Focal Vibration Tool on the Biomechanics of the Lower Limb
Brief Title: To Assess the Efficacy of a Localized Focal Vibration Tool on the Muscular Response to Five Countermovement Jumps in Healthy Soccer Players
Acronym: EVIFOBIOMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Rovira i Virgili (Other)
Responsible Party: Principal Investigator, Gisela Cisa Ribas, Physiotherapist, University Rovira i Virgili
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 195/2021
Record Dates: First submitted 2025-04-09; First posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Prevention and Control; Healthy People Programs
Keywords: vibration; biomechanics; lower extremity; football; plyometric exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Active Comparator): The intervention group performed a 20-minute warm-up divided into four equal parts. First, they performed lower limb joint mobility exercises, followed by pedaling a stationary bicycle at 60-70 rpm. They then performed specific plyometric exercises for jumping and 8 minutes of active rest.
  After completing the warm-up, the subjects performed five countermovement jumps. They were then fitted with focal vibration devices with the heads set at 120 Hz, while they pedaled for 10 minutes at 90-100 rpm. Once the time was up, they performed the five countermovement jumps again.
  The protocol was identical for all three days of the intervention.
  Interventions: Other: Non invasive focal vibration with heads
- Placebo group (Placebo Comparator): The placebo group performed a 20-minute warm-up divided into four equal parts. They first performed lower limb joint mobility exercises, followed by pedaling a stationary bicycle at 70-80 rpm. They then performed specific plyometric exercises for jumping and 8 minutes of active rest.
  After completing the warm-up, the subjects performed five countermovement jumps. They were then fitted with the focal vibration devices without the headpieces, so as not to produce any tactile stimulation, at 0 Hz, while they pedaled for 10 minutes at 90-100 rpm. Once the time was up, they performed the five countermovement jumps again.
  The protocol was identical for all three days of the intervention.
  Interventions: Other: Non invasive focal vibration without heads

INTERVENTIONS:
Other: Non invasive focal vibration with heads — 3 sessions over 3 consecutive weeks, with one intervention day per week. Non invasive focal vibration at 120 Hz for 10 minutes while pedaling at 90-100 rpm
  Arms: Intervention group
Other: Non invasive focal vibration without heads — 3 sessions over 3 consecutive weeks, with one intervention day per week. Non invasive focal vibration at 0 Hz for 10 minutes while pedaling at 90-100 rpm
  Arms: Placebo group

SUMMARY:
This research study aims to introduce the localized focal vibration tool. To this end, a 3-week protocol with a single session per week was created.

In the one hand, the study subject must be a soccer player, regardless of whether male or female, and must not be suffering from any active injury.

All subjects must complete an identical warm-up before beginning the noninvasive intervention using the vibration tool.

The warm-up consists of various joint mobility exercises for the legs, a brief cardio session by pedaling a stationary bicycle, and finally, jumping exercises to properly activate the main muscles of the lower limbs and thus be able to begin the intervention protocol.

In the other hand, the study subjects are divided into two groups: intervention and placebo.

Neither the study subject nor the research team knows who belongs to each group; only the person handling the focal vibration tool will know.

To begin the intervention, three surface electromyography probes are placed on the vastus medialis of the quadriceps, the tibialis anterior, and the internal gastrocnemius, and the subject is asked to perform five countermovement jumps barefoot and without moving their arms to gain momentum.

The subject then pedals at 90-100 rpm on a stationary bicycle while wearing the sensors of the 120 Hz focal vibration tool for 10 minutes.

The intervention group wears headgear to ensure tactile stimulation, while the placebo group does not wear headgear, thus ensuring that there is no tactile stimulation.

After the pedaling period, the electromyography sensors are reapplied to the lower limb in the anatomical areas described above, and the same jumping protocol is followed again.

This intervention is identical for the 3 days of recording.

This noninvasive intervention protocol aims to demonstrate the effectiveness of the 120 Hz focal vibration tool in recruiting muscle fibers in the targeted muscles through numerical improvements in muscle electrical activity and improved countermovement jump parameters.

A three-day follow-up period was established to determine when any improvement from the application of focal vibration therapy begins.

All study subjects are volunteers to participate during the official soccer season for their respective age group and may withdraw from the study at any time if they wish.

ELIGIBILITY:
Inclusion Criteria:

* Practice soccer at least three times a week.
* Do not suffer from any alterations or pathologies prior to or during the study in the area of interest for the research.

Exclusion Criteria:

* Having a lower limb disorder or pathology
* Receiving any type of lower limb treatment from a healthcare professional or receiving pseudoscientific treatments.
* Having any absolute or relative contraindications to measurement tests, surface electromyography, inertial sensor, and/or focal vibration.
* Refuse to sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-01-02 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Heigh of countermovement jump with G-sensor | From enrollment to the end of treatment at 3 weeks"
  Average height of the second sacral vertebra difference of the 5 countermovement jumps over the 3 days of intervention. This difference is evaluated using the inertial G sensor on the second sacral vertebra. It is a device that is placed on the subject's waist, secured with a belt, in order to measure the difference in jump height in centimeters.

SECONDARY OUTCOMES:
Muscle electrical activity with surface electromyography | From enrollment to the end of treatment at 3 weeks"
  The difference in muscle electrical activation of the following muscles is evaluated: Vastus medialis of the quadriceps, Tibialis anterior and Gastrocnemius medialis, of the dominant lower extremity in the five countermovement jumps over the 3 days of intervention. The electromyographic values, in millivolts, are obtained using the FREEMG 1000 tool.
Velocity of countermovement jump with G-sensor | From enrollment to the end of treatment at 3 weeks"
  Average velocity of the second sacral vertebra difference of the 5 countermovement jumps over the 3 days of intervention. This difference is evaluated using the inertial G sensor. It is a device that is placed on the subject's waist, secured with a belt, in order to measure the difference values of the velocity in meters/seconds.
Power of countermovement jump with G-sensor | From enrollment to the end of treatment at 3 weeks"
  Average to power difference of the 5 countermovement jumps over the 3 days of intervention. This difference is evaluated using the inertial G sensor on the second sacral vertebra. It is a device that is placed on the subject's waist, secured with a belt, in order to measure the difference values of the power in Watts.

CONTACTS AND LOCATIONS:
Locations (1):
- Rovira i Virgili University, Reus, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li W, Li C, Xiang Y, Ji L, Hu H, Liu Y. Study of the activation in sensorimotor cortex and topological properties of functional brain network following focal vibration on healthy subjects and subacute stroke patients: An EEG study. Brain Res. 2019 Nov 1;1722:146338. doi: 10.1016/j.brainres.2019.146338. Epub 2019 Jul 16. PMID 31323197
- [Background] Brunetti O, Botti FM, Brunetti A, Biscarini A, Scarponi AM, Filippi GM, Pettorossi VE. Effects of focal vibration on bone mineral density and motor performance of postmenopausal osteoporotic women. J Sports Med Phys Fitness. 2015 Jan-Feb;55(1-2):118-27. PMID 25642687
- [Background] Murillo N, Valls-Sole J, Vidal J, Opisso E, Medina J, Kumru H. Focal vibration in neurorehabilitation. Eur J Phys Rehabil Med. 2014 Apr;50(2):231-42. PMID 24842220